CLINICAL TRIAL: NCT00327561
Title: Effects of Non-Surgical Periodontal Therapy on Endothelial Function A Randomized Controlled Clinical Trial
Brief Title: Effect of Intensive Periodontal Therapy on Vascular Function
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastman Dental Insitute and Hospital (Other)
Collaborators: University College London Hospitals (Other); British Heart Foundation (Other); The European Research Group on Periodontology (ERGOPerio) (Network); Johnson & Johnson (Industry); CORDA, The Heart Charity (Other); European Social Fund (Other); Italian Society of Periodontology (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCLH03/E007
Record Dates: First submitted 2006-05-16; First posted 2006-05-18 (Estimated); Last update posted 2006-05-18 (Estimated); Status verified 2005-03

CONDITIONS: Periodontitis
Keywords: Inflammation; Periodontitis; Endothelial function; Atherosclerosis; Controlled trial
MeSH Terms: conditions — Periodontitis; Inflammation; Atherosclerosis

INTERVENTIONS:
Procedure: Intensive periodontal therapy
Procedure: Community based periodontal therapy

SUMMARY:
The hypothesis of the existence of a causal association between the systemic infectious/inflammatory burden represented by periodontitis and endothelial function assessed by flow mediated dilatation of the brachial artery (FMD) is the subject of the proposed investigation.

The objective of this randomized controlled clinical trial is to evaluate the effects of periodontal therapy on endothelial function assessed by Flow mediated dilatation (FMD).

The rationale for this project is twofold:

* Establish the extent of acute systemic inflammation and endothelial dysfunction associated with the delivery of subgingival instrumentation for the treatment of chronic periodontitis
* Establish whether or not improved control of chronic periodontal infections results in improved endothelial function and thus the existence of a causal association between periodontitis and endothelial dysfunction.

DETAILED DESCRIPTION:
In the last decade considerable evidence has supported the hypothesis that chronic low-grade infections, periodontitis included, and the inflammatory responses associated with them may play a significant role in the onset of atherosclerosis. An inflammatory alteration of the normal endothelial activity is thought to be one of the mechanisms that may link infection with atherosclerosis. It consists of loss of the normal vasodilation, antiplatelet and antithrombotic properties of the vascular walls and it is frequently called endothelial dysfunction. Impaired endothelium-dependent dilatation, an early functional marker of endothelial dysfunction has been demonstrated in young populations with family history of cardiovascular diseases. In the past 15 years a new non invasive and reproducible technique called Flow mediated dilatation (FMD) has been used to assess endothelial function.

Periodontitis is a chronic infection of the tooth supporting apparatus caused primarily by anaerobic gram negative bacteria organised in a biofilm (commonly known as sub-gingival dental plaque); it leads to inflammatory destruction of the periodontal ligament and alveolar bone and eventually to tooth exfoliation. Periodontitis is highly prevalent in both industrialised and developing countries with 10-15% of the adult population being affected by severe forms of this disease. Recognized risk factors include genetic polymorphisms in inflammatory genes, environmental exposures such as cigarette smoking, and systemic diseases such as diabetes. Local periodontal production of prostaglandins and pro-inflammatory cytokines has been associated with activation of matrix metalloproteinases and eventually to destruction of the periodontal ligament and alveolar bone. It is the primary cause of tooth loss in adult populations and as such leads to long term disability and increased treatment needs.

Local periodontal infections have been associated with a systemic response characterized by increased serum levels of C-reactive protein (CRP), hyper-fibrinogenemia, moderate leukocytosis, as well as increased serum levels of IL-1 and IL-6 when compared with unaffected control populations.

Several epidemiological studies have associated increased levels of acute phase markers with higher risk for cardiovascular atherosclerotic events. Among these markers, C-reactive protein is considered to be one of the most sensitive and probably to be an independent risk factor of atherosclerosis. It is produced by the liver presumably for adaptive or defensive reasons in response to a variety of inflammatory stimuli, including chronic low grade infections.

In a recently completed pilot trial we have been able to establish that treatment of periodontal infections resulted in a significant decrease in serum CRP. In that study, treatment of periodontal infections led to a significant decrease in serum CRP (0.5 mg/L, 95% CI 0.4 to 0.7 mg/L) and IL6 in otherwise healthy individuals affected with severe, generalized periodontitis and indicated that periodontitis contributed to the systemic inflammatory responses.

The treatment associated decrease in systemic inflammatory markers observed in this study supports the hypothesis that periodontal infections, along with chronic low grade infections in other body districts, contribute to the inflammatory burden of an individual and may play a contributory etiologic role in atherosclerosis. It remains to be established whether or not the observed improvements in serum CRP have an impact on functional vascular parameters and endothelial function/dysfunction.

The relationship between periodontal treatment and changes in serum CRP is likely to be bimodal: an increase associated with the delivery of the standard subgingival instrumentation and the associated bacteremia and tissue damage is expected shortly after treatment is delivered.

Preliminary trials from our group aimed at the establishment of the pattern of CRP changes in the first days following delivery of periodontal therapy. The data indicate that serum CRP levels sharply increase after treatment but that values tend to return to baseline levels by one week. This bimodal pattern of changes in serum CRP levels is important since previous investigations have established links between functional vascular parameters such as flow mediated dilatation (FMD) and serum markers of systemic inflammation such as CRP.

Periodontal therapy therefore may lead to an initial improve FMD parameters in subject were periodontitis contributes to systemic inflammation and atherosclerosis. The hypothesis of the existence of a causal association between the systemic infectious/inflammatory burden represented by periodontitis and endothelial function assessed by FMD is the subject of the proposed investigation.

Compare the effects of an intensive periodontal treatment regimen with a community based periodontal care approach in terms of changes in:

* Flow mediated dilatation of the brachial artery (primary outcome)
* Acute phase response in serum (CRP, IL-6,fibrinogen)
* Clinical periodontal parameters: PI, BoP, PPD (CAL)
* Presence of periodontal pathogens in the periodontal pockets before and after treatment
* Patient perception and adverse events associated with the treatment experience This will be a randomized controlled clinical trial. Its design will be parallel arm, single blind; outcomes will be evaluated over a 6 months period and will include approximately 120 subjects. Two interventions will be compared: test treatment will be an intensive regimen of periodontal therapy consisting of oral hygiene instructions and subgingival debridement delivered at two appointments over a 24 hour period; control treatment will consist of a community based periodontal care approach consisting of supragingival removal of deposits delivered at two appointments over a 24 hour period. The control group will receive the intensive regimen upon completion of the study or upon evidence that periodontitis is progressing. Subjects with moderate to severe periodontitis will be recruited among those referred for care to the Periodontal Clinic of the Eastman Dental Hospital. The primary outcome measure of this study will be changes in Flow Mediated Dilatation (FMD) of the brachial artery. Secondary outcomes will include changes in serum CRP and plasma fibrinogen. Periodontal, microbiological and subjective outcomes will be evaluated as control outcomes. The primary and the secondary outcome variables will be evaluated before treatment and at 1 day, 7 days, 2 months and 6 months following completion of treatment. Subjects will be randomized to treatment stratifying for smoking status by a study registrar. Treatment allocation will be concealed to study personnel by using opaque envelopes and to the examiner by making treatment records unavailable. All laboratory and FMD analyses will be performed by unrelated study personnel blind with respect to treatment allocation or stage of progression of the trial. Intent to treat analyses will be performed by a statistician blind with respect to treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 35 and 60 and in good general health.
* Ability and willingness to follow study procedures and instructions.
* Must have read, understood and signed the Informed Consent.
* Must have generalized, moderate to advanced chronic periodontitis.
* 40-100 pockets with a PD of > 5 must bleed on probing.
* Absence of other significant oral infections.

Exclusion Criteria:

* Pregnant or lactating females or females of child bearing potential not using acceptable methods of birth control (hormonal, barriers or abstinence).
* Patients chronically treated (i.e., two weeks or more) with any vasoactive medication (i.e., antihypertensive) or lipid lowering therapy.
* Patients who started taking nonsteroidal anti-inflammatory drugs within two months prior to the baseline visit.
* Diagnosis of uncontrolled metabolic diseases including diabetes, kidney, liver, or cardiovascular diseases.
* Use of systemic antibiotics in the preceding 3 month.
* Patients taking steroid medications except for acute topical treatment.
* Patients with active infectious diseases such as hepatitis, HIV, or TB.
* Patients who require antibiotic pre-medication for the performance of periodontal examination or treatment.
* Patients who received a course of periodontal treatment within the last 6 months.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120
Dates: Start 2003-09; Study Completion 2005-03

PRIMARY OUTCOMES:
Flow mediated dilatation of the brachial artery

SECONDARY OUTCOMES:
Serum inflammatory and endothelial function markers

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Tonetti, DMD PhD, Principal Investigator — University College London Hospitals and University of Connecticut Health Center
Locations (2):
- United Kingdom (2):
  - UCL Eastman Dental Institute and Hospital, London
  - UCL Vascular Biology Laboratory - Great Ormond Street Hospital, London

REFERENCES:
- [Background] D'Aiuto F, Parkar M, Nibali L, Suvan J, Lessem J, Tonetti MS. Periodontal infections cause changes in traditional and novel cardiovascular risk factors: results from a randomized controlled clinical trial. Am Heart J. 2006 May;151(5):977-84. doi: 10.1016/j.ahj.2005.06.018. PMID 16644317
- [Background] D'Aiuto F, Nibali L, Parkar M, Suvan J, Tonetti MS. Short-term effects of intensive periodontal therapy on serum inflammatory markers and cholesterol. J Dent Res. 2005 Mar;84(3):269-73. doi: 10.1177/154405910508400312. PMID 15723869
- [Background] D'Aiuto F, Parkar M, Andreou G, Suvan J, Brett PM, Ready D, Tonetti MS. Periodontitis and systemic inflammation: control of the local infection is associated with a reduction in serum inflammatory markers. J Dent Res. 2004 Feb;83(2):156-60. doi: 10.1177/154405910408300214. PMID 14742655
- [Background] D'Aiuto F, Tonetti MS. Contribution of periodontal therapy on individual cardiovascular risk assessment. Arch Intern Med. 2005 Sep 12;165(16):1920-1. doi: 10.1001/archinte.165.16.1920. No abstract available. PMID 16157839
- [Background] D'Aiuto F, Parkar M, Brett PM, Ready D, Tonetti MS. Gene polymorphisms in pro-inflammatory cytokines are associated with systemic inflammation in patients with severe periodontal infections. Cytokine. 2004 Oct 7;28(1):29-34. doi: 10.1016/j.cyto.2004.06.005. PMID 15341923
- [Background] D'Aiuto F, Parkar M, Tonetti MS. Periodontal therapy: a novel acute inflammatory model. Inflamm Res. 2005 Oct;54(10):412-4. doi: 10.1007/s00011-005-1375-4. PMID 16283108
- [Background] D'Aiuto F, Parkar M, Andreou G, Brett PM, Ready D, Tonetti MS. Periodontitis and atherogenesis: causal association or simple coincidence? J Clin Periodontol. 2004 May;31(5):402-11. doi: 10.1111/j.1600-051X.2004.00580.x. PMID 15086624